CLINICAL TRIAL: NCT06294366
Title: Bipolar Transurethral Enucleation Versus Resection in the Treatment of Benign Prostatic Hyperplasia: a Comparative Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Menoufia University (Other)
Responsible Party: Principal Investigator, Mohamed Abdelgawad Rokba, Assistant lecturer, Urology department, Faculty of Medicine, Menoufia University, Menoufia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MenoufiaU2022
Record Dates: First submitted 2024-01-02; First posted 2024-03-05 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Prostatic Hyperplasia; Prostate Enucleation
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Bipolar enucleation (Active Comparator): Bipolar enucleation of the prostate larger than 60 gm
  Interventions: Device: Bipolar Bowa device
- Bipolar TURP (Active Comparator): Bipolar transurethral resection of the prostate larger than 60 gm
  Interventions: Device: Bipolar Bowa device

INTERVENTIONS:
Device: Bipolar Bowa device — Bipolar Bowa device used in prostatic resection and enucleation

SUMMARY:
Benign prostatic hyperplasia (BPH) is a common chronic progressive disease resulting in the enlargement of the prostate gland and bladder outlet obstruction in aging men .

Because of the increasing aged population and advancements in diagnostic tools, the incidence and importance of BPH have increased . BPH can be treated either with watchful waiting, drug therapy, or surgery being the most effective treatment option for BPH .

Transurethral resection of the prostate (TURP) has been recognized as the standard treatment for BPH with morbidity rate varies from 18% and 26% Until now, only open prostatectomy and transurethral Holmium laser enucleation of the prostate (HoLEP) have shown an equal efficacy and durability compared to TURP

DETAILED DESCRIPTION:
Benign prostatic hyperplasia (BPH) is a common chronic progressive disease resulting in the enlargement of the prostate gland and bladder outlet obstruction in aging men.

Because of the increasing aged population and advancements in diagnostic tools, the incidence and importance of BPH have increased. BPH can be treated either with watchful waiting, drug therapy, or surgery being the most effective treatment option for BPH.

Transurethral resection of the prostate (TURP) has been recognized as the standard treatment for BPH with morbidity rate varies from 18% and 26%.

Until now, only open prostatectomy and transurethral Holmium laser enucleation of the prostate (HoLEP) have shown an equal efficacy and durability compared to TURP.

An increasing number of endoscopic techniques have been attempted to overcome these complications. One of the technical modifications of TURP is the bipolar transurethral resection of the prostate (B-TURP) which enables urologists to use normal saline solution as an irrigation fluid to overcome the risk of TUR syndrome occurrence and requires less energy.

Currently bipolar TURP is considered a valid alternative to monopolar TURP offering similar efficacy with lower peri-operative morbidity.

Moreover, the bipolar system can also be used to enucleate entire large prostate glands, achieving an effective alternative to TURP and open simple prostatectomy (OP), and reducing complications associated with these techniques, including risk of bleeding and blood transfusion.

The crux of the idea behind enucleation is that it depends on removing the prostatic tissue along the surgical capsule as in open prostatectomy, but in a minimally invasive setting, with the same tissue removal capability.

Despite a growing amount of data reported in the literature, it remains unclear how PKEP compares to more established B-TURP in the surgical treatment of BPH

The aim of the study is to assess the surgical efficacy, safety, and peri-operative morbidity of bipolar plasmakinetic enucleation of the prostate (PKEP) in comparison with bipolar transurethral resection of the prostate (B-TURP) for the treatment of patients with symptomatizing prostates.

A prospective randomized controlled study was conducted in 52 patients diagnosed with lower urinary tract symptoms due to benign prostatic hyperplasia (BPH) whose prostates > 60 gm. The perioperative parameters, therapeutic effects and complications were compared between the two groups before and 3 months after surgery.

Preoperative evaluation included detailed medical history, thorough clinical examination, International Prostate Symptom Score (IPSS), digital rectal examination (DRE), prostate volume, post-voiding residual urinary volume (PVR), PSA level and maximum flow rate (Qmax).

Intraoperative evaluation included operative time, irrigating fluid volume, the volume of removed prostate tissue, blood loss, and intraoperative complications.

Postoperative evaluation included the mean hemoglobin and hematocrit differences, catheterization period, hospital stay, postoperative complications and follow up IPSS, PVR and Qmax.

ELIGIBILITY:
Inclusion Criteria:

* all patients with symptomatizing BPH who have a prostate volume > 60 gm and indicated for surgical treatment.

Exclusion Criteria:

* patients with small fibrotic prostates, high PSA (not co-inciding with BPH), neurogenic bladder.

Ages: 50 Years to 90 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2022-06-12 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-10-30 (Actual)

PRIMARY OUTCOMES:
Assessing and comparing the safety, the surgical efficacy and peri-operative morbidity of bipolar enucleation of the prostate and bipolar transurethral resection of the prostate for the treatment of patients with symptomatizing prostates. | one year
  Preoperative evaluation will include detailed medical history, thorough clinical examination, international prostate symptom score (IPSS), digital rectal examination (DRE), prostate specific antigen [Prostatic specific antigen (free/total)], maximum flow rate (Qmax), and pelvi-abdominal ultrasound to assess prostate size and post-voiding residual urinary volume (PVR).
  Intraoperative evaluation will include operative time, irrigating fluid volume, the volume of removed prostate tissue, and intraoperative complications.
  Postoperative evaluation will include the mean haemoglobin difference, hematocrit level, catheterization period, hospital stay, medications, analgesics, and follow up maximum flow rate (Qmax).

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of medicine, Shibīn al Kawm, Menoufia, Egypt